CLINICAL TRIAL: NCT04351620
Title: High-dose Hydroxychloroquine for the Treatment of Ambulatory Patients With Mild COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB20-0572
Record Dates: First submitted 2020-04-14; First posted 2020-04-17 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
Keywords: hydroxychloroquine
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hydroxychloroquine (Experimental): Hydroxychloroquine 1200 mg daily administered as 600 mg BID for five days or until fevers abate (maximum ten days of treatment allowed).
  If patients report gastrointestinal discomfort, the dose will be administered as 400 mg TID.
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine — Tolerability study of HCQ 1200 mg administered daily in divided doses for a duration of 5-10 days

SUMMARY:
This study aims to examine the tolerability of high dose hydroxychloroquine in patients with COVID-19 who are not yet hospitalized, but have risk factors for disease progression and complications.

DETAILED DESCRIPTION:
This is a single arm and single-center tolerability study of high dose HCQ therapy in outpatient adult participants with mild COVID-19. In vitro studies have shown antiviral effects of HCQ against SARS Cov-2, but the clinical outcomes in the disease have been variable. The hypothesis is that targeting high risk patients earlier in the disease course and with a higher dose regimen are both required to see improvement in disease outcome measures in COVID-19. This study aims to prove the tolerability of high dose HCQ in this setting.

Patients are selected based on the identification of risk factors associated with more severe disease outcomes. Investigators will enroll twenty patients and perform a detailed Tele-health interview to ensure they meet eligibility criteria and provide informed consent. 1200 mg hydroxychloroquine daily will be prescribed, in divided doses.The subjects will be required to monitor their temperatures twice daily and a daily telephone call with an investigator will review symptoms of disease and potential side effects of the drug. Subjects can discontinue the medication after five days if they no longer have fever, or take the medication for up to ten days if required for fever resolution.

ELIGIBILITY:
Inclusion Criteria:

* Being tested positive for SARS-Cov-2 in outpatient setting in drive-thru, ED, or ambulatory clinics at the University of Chicago within 72 hours of enrollment.
* Age >18
* Fever >100.4 F by any conventional clinical method (forehead, tympanic, oral, axillary, rectal) within 48h prior to enrollment
* Mild COVID-19, defined as the presence of any symptom consistent with an upper respiratory tract infection, including dry cough, sore throat, nasal congestion, fatigue, myalgia, headaches.

Subjects must meet all the above-mentioned criteria, in addition to at least one of the following criteria:

* Age > 55
* Pre-existing pulmonary disease: airway diseases (asthma, chronic obstructive pulmonary disease, bronchiectasis, cystic fibrosis), history of active or treated lung cancer, history of pneumectomy, interstitial lung diseases, pulmonary hypertension, sleep apnea.
* Diabetes: uncontrolled or controlled diabetes
* Hypertension
* Chronic kidney disease stage 1-3
* History of cardiovascular disease with an electrocardiogram available to the physician-investigator through the subject's electronical medical record within the past thirty days showing a normal QT interval (QT < 500 ms).
* History of immunosuppression
* Active cancer diagnosis, on palliative treatment or requiring current therapy with antimetabolic agents, immunotherapy or radiotherapy.
* At least one fever every 24 hours for > 72h

Exclusion Criteria:

* Participation in any other clinical trial of an experimental agent treatment for COVID-19
* Current hospitalization
* Known hypersensitivity to hydroxyxhloroquine or chloroquine
* Known chronic kidney disease, stage 4-5, or receiving dialysis
* History of retinal disease
* History of uncontrolled hypertension, defined as systolic blood pressure > 180 mmHg and or diastolic blood pressure > 100 mmHg at the most recent physical medical encounter or by patient report.
* History of QT prolongation (QT > 500 ms) or history of Torsades de Pointes
* History of arrhythmias
* Current use of loop diuretics and potassium supplementation or documented history of hypokalemia.
* Pregnancy and lactation
* Known glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Current use of any of the following medications: flecainide (Tambocor), amiodarone (Cordarone, Pacerone), digoxin (Digox, Digitek), procainamide (Procan, Procanbid), propafenone (Rythmal), antiepileptic agents (phenytoin, phenobarbital, valproic acid, lamotrigine, topiramate), tamoxifen, tricyclic antidepressants (nortriptyline, amitriptyline, imipramine, clomipramine)
* Inability to monitor body temperature (oral, axillary, tympanic or frontal) at least twice a day from study enrollment day (Day 1) to the end of the study (Day 14).
* Inability to provide informed consent to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Tolerability of high dose HCQ as measured by HCQ dose modification and ability to complete course | 14 days
  Number of subjects requiring HCQ dose modifications
Tolerability of high dose HCQ as measured by discontinuation of HCQ before end of course | 14 days
  Number of subjects that discontinue HCQ
Tolerability of High Dose HCQ as measured by Adverse Events | 14 days
  Number of Adverse Events observed in all subjects for the duration of the study

SECONDARY OUTCOMES:
Rate of hospitalization due to COVID-19 as measured by number of patients hospitalized | 14 days
  Number of patients admitted to hospital during study period
Time to defervescence as measured in days while on treatment protocol | 14 days
  The number of days to reach first fever normalization (criteria for normalization: temperature < 100.4 F)
Resolution of other COVID-19 symptoms measured in days while on treatment protocol | 14 days
  Number of days to resolve other symptoms, as assessed by a standardized questionnaire for symptom assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Reem Jan, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided